CLINICAL TRIAL: NCT05977660
Title: Cross-cultural Adaptation and Cut-off Score Determination of the Turkish Version of the Cumberland Ankle Instability Tool (CAIT-TR)
Brief Title: Turkish Language and Cross-cultural Adaptation of the Cumberland Ankle Instability Tool
Acronym: CAIT-TR
Status: Completed | Type: Observational
Sponsor: Eskisehir Technical University (Other)
Responsible Party: Principal Investigator, Celil Kaçoğlu, Associated profesor, Eskisehir Technical University
Other Study IDs: EskisehirTU-SBF-CK-01
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ankle Injuries; Instability, Joint
Keywords: ankle instability; chronic ankle instability; cumberland ankle instability tool; cross-cultural adaptation; validity and reliability; self-reported questionnaire; CAIT; Turkish language and cultural adaptation
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With chronic ankle instability (CAI): Participations with CAI diagnosed by a medical doctor
  Interventions: Diagnostic Test: Cumberland ankle instability tool for diagnose to determine ankle instability and its severity
- control (without CAI): Participations without CAI who didn't have any ankle injury 2 years before the study recruitment
  Interventions: Diagnostic Test: Cumberland ankle instability tool for diagnose to determine ankle instability and its severity

INTERVENTIONS:
Diagnostic Test: Cumberland ankle instability tool for diagnose to determine ankle instability and its severity — CAIT is a Patient-reported measures of outcome (PROM) and it is very simple, reliable, and valid measurement tool that is used without comparing with the contralateral ankle, which consists of 9 questions and is scored between 0 and 30, developed by Hiller and her colleagues in 2006 to measure the severity of functional ankle instability. Low scores of the participants indicate poor ankle stability, while high scores indicate good ankle stability.

SUMMARY:
Cumberland Ankle Instability Tool (CAIT) is a valid patient-reported outcome measure (PROM) to determine the presence of ankle instability (AI) and assess its severity. The aim of current study is to adapt the CAIT into the Turkish language, test its psychometric properties and determine cut-off score in the Turkish population with AI compare to healthy counterparts. In order to evaluate the Turkish version of CAIT (CAIT-TR), data will obtaine from 200-250 participants with and without AI. Test-retest reliability, internal consistency, cut-off score, and ceiling and floor effects will evaluate.

DETAILED DESCRIPTION:
The foot and ankle are the most common injured body parts after the knee in the general population and athletes. Ankle sprain, which is the most common injury in the ankle, consists of more than 80% of all ankle injuries. While the rate of ankle injury among all sports injuries is 23%, according to a study, the most common sports injury seen among 33 sports is ankle sprain (76.7%). Taking into account that ankle sprains are considered insignificant by athletes and coaches and that 40-55% of individuals who experienced ankle sprains for the first time do not seek medical support and treatment from a healthcare professional, it is understood that this rate is higher than it seems. Almost half of the ankle sprains (49.3%) occur during athletic activities, and these ankle sprains that are related to athletic activity are mostly common in basketball (41.1%), football (9.3%), and soccer (7.9%). The incidence of ankle sprain is seen higher in the field (i.e. field, court) and team sports (such as rugby, soccer, volleyball, handball, basketball, American football, Australian football, Gaelic football, tennis, netball, lacrosse, and field hockey). The incidence of ankle sprains, which is quite common in athletes and also in the general population, has been seen as higher in women compared to men, in adults compared to adolescents, and in children compared to adolescents.

Despite the acute symptoms of ankle sprain disappearing very quickly, most individuals develop long-term symptoms such as pain, a feeling of instability, a perception of weakness, and crepitus, which play a role in the development of chronic ankle instability (CAI) after the injury. Seventy-four percent of individuals with an ankle sprain show at least one symptom for 1.5-4 years following the injury, and 32% of individuals with a history of ankle sprain have chronic complaints even 7 years after the injury. One of the most common of these permanent problems is CAI and the feeling of "giving way", which occurs as a result of multiple recurrences of ankle sprain. Ankle stabilization is an integral part of normal movement and minimizes the risk of ankle sprain during sports activities.

Ankle sprains have a high recurrence rate, and approximately 30% of individuals with a history of ankle sprains experience CAI. CAI is observed within 1 year after the injury in 40.5% of individuals who have had their first ankle sprain, and the incidence of CAI can reach up to 70% shortly after the sprain. The chronicity of recurrent sprains, the decrease in physical activity level and quality of life, the increase in post-traumatic ankle osteoarthritis rates, and the large financial costs cause deterioration in the athletic performance of athletes. Considering all these results, the necessity of an appropriate approach to prevent injury and comprehensive rehabilitation programs is a fact.

Although there are different definitions such as chronic ankle instability, functional ankle instability, and mechanical ankle instability. The term CAI is most frequently used when describing patients who report that their symptoms continue after their first ankle sprain, and the most reported losses associated with CAI are the number/repeat of sprains and the sensation of giving way in the ankle joint. Ankle instability is a common clinical problem in athletes, in which various complex mechanical and neuromuscular factors play a role. Two hypothetical causes of CAI are defined as mechanical instability and functional instability. Mechanical instability (MI) is defined as ankle movement beyond the physiological limits of the ankle range of motion. The term laxity is often used synonymously with mechanical instability. Functional instability (FI) is defined as ankle instability due to proprioceptive and neuromuscular deficits or the subjective feeling of recurrent and symptomatic ankle sprains (or both). As it can be understood from here, the perception of individuals is an important issue in CAI diagnoses.

Interventions by clinicians and physiotherapists are usually standard medical tests and practices and their evaluations, which initially provide key information based on various screening methods, joint range of motion, and joint and tissue stability. With these results, which do not include the perspective of the individual, in addition to the measurable characteristics of the individual, it is largely incomprehensible how the patient feels about his health status. The goal of most healthcare services is to improve patient's well-being, and patients themselves are probably the ones who can best assess their feelings. Patient-reported measures of outcome (PROM) convert qualitative entities such as anxiety, pain, or social functioning that cannot be directly observed, or that are impractical or impossible to directly observe (for example, the performance of daily activities), into quantitative scores that can be processed mathematical statements such as patient perceptions of certain aspects of their own health. PROMs can provide both valid and reliable results that directly reflect the patient's own perspective, without the interpretation of the doctor or others, in response to a series of questions asked about patients' views and priorities regarding the treatment they receive or their own health status, how they feel, their quality of life, or their functional status. They are questionnaire-like scales that were developed to measure patients' own assessments of their health and health-related quality of life. PROMs such as the Western Ontario Shoulder Instability Index (WOSI) for shoulder instability, knee injury, osteoarthritis outcome score (KOOS) for knee problems, and Victorian Sports Assessment Institute (VISA) for tendinopathies are widely used in sports health. PROMs, which are useful clinical tools to obtain information about the perceived health status of patients, are becoming increasingly popular for clinicians to measure the changes in patient's health status over time. PROMs are usually general, regional, or disease-specific. While using scales such as the SF-36 health questionnaire in the general evaluation of health status, regional scales designed to be sensitive to the characteristics of the population to assess problems and functions specific to certain regions of the musculoskeletal system, such as general shoulder, arm and hand disorders (DASH), Victorian sports institute for Achilles assessment (VISA-A) or condition-specific examples such as patellar tendinopathy (VISA-P). Disease-specific rating scales are designed to assess function, pain, and problems in specific conditions. Scales whose reliability, validity, and responsiveness have been scientifically tested are the most useful scales.

A common reason for translating and adapting PROMs from one language to another is that there is an absence of a local language-adapted version of a specific PROM required for clinical or academic research. If a PROM has been developed using valid methods with data from relevant patient groups, and there is content relevance and scope for patients, it is a better reason to translate and adapt an existing PROM than to develop a new PROM. This method is both easier and less time-consuming. Adapting a PROM to a new language or culture is important. Even for languages spoken by many people globally in different countries, such as Spanish, English, and Arabic, there can be quite many versions of the same base language, as the habits and cultures of different countries can differ significantly. The same word or phrase may have different connotations and meanings in different countries, or objects may be described by different words in the same language, depending on culture or geography. Also, living conditions can be very different in language areas depending on socioeconomic, religious, and cultural conditions that often vary between countries. Therefore, the content of items in a PROM may not have the same meaning or precaution when translated into a new culture.

Some PROMs are used by clinicians and researchers to evaluate the effects of treatment interventions for individuals with foot and ankle pathological conditions and subsequent disorders. Although there are at least 17 PROMs commonly used to evaluate patients with ankle instability in the literature, only 3 of them were developed by including patients (Cumberland ankle instability, Lower extremity function scale, Foot and ankle ability measure) and Cumberland Ankle Instability Tool (CAIT), which is one of these scales with the best internal consistency and best psychometric properties can be used to diagnose instability as well as an assessment tool.

CAIT is a very simple, reliable, and valid measurement tool that is used without comparing with the contralateral ankle, which consists of 9 questions and is scored between 0 and 30, developed by Hiller and her colleagues in 2006 to measure the severity of functional ankle instability. Low scores of the participants indicate poor ankle stability, while high scores indicate good ankle stability. The International Ankle Consortium (IAC) considers that patient-reported instability should be measured with valid questionnaires and recommends using CAIT ≤24 scores as a cut-off value for inclusion criteria. Different cut-off scores have been revealed in various studies conducted in different groups and cultures. For example, although it is stated that ≥ 28 scores indicate stability and ≤ 23 scores indicate instability, Hiller et al. calculated the cut-off score as 27.5. In recent study cut-off score was calculated as ≤25. Another study conducted on the athlete population, it is stated that those who score above 28 are unlikely to have AI, while individuals who score ≤27 are likely to have AI.

The fact that the original language is English limits CAIT's use of this tool in ankle instability assessments of many non-English speaking countries and communities around the world. Testing the psychometric properties of CAIT, which is reliable and valid for English language and culture. In different languages and cultures, is very important to popularize the use of this measurement tool. CAIT has been translated from the original language English to many languages such as Spanish, Brazilian-Portuguese, Korean, Japanese, Dutch, Persian, French, Cantonese, Taiwanese, Arabic, Thai, Greek, and Urdu. Besides all these, there is also a digital version of CAIT .

There are some foot and ankle-specific scales such as the Identification of Functional Ankle Instability (IdFAI), the Olerud-Molander Ankle Score (OMAS), Foot and Ankle Ability Measure (FAAM), Foot and Ankle Outcome Score, Self-Reported Foot and Ankle Score which have been adapted to the Turkish population and language and tested for reliability and validity.

Since there is no Turkish version of CAIT, it cannot be used by researchers and clinicians working with Turkish-speaking population to determine ankle instability and severity. Considering that the demand for such PROM scales, which have widespread applicability to be used in both clinical and scientific research, is increasing, the aim of the current study is to adapt CAIT from its original language to Turkish (CAIT-TR) and Turkish culture and examine its psychometric properties in participants with and without AI.

ELIGIBILITY:
Inclusion Criteria:

* Participants consisted of women and men aged between 18 and 35.
* The volunteers to be included in the study are male and female individuals who have a history of ankle instabililty in the last two months at least for the study group and healthy individuals without any injury and the selection will be made at randomly.

Exclusion Criteria:

* As criteria for excluding the participants in the study; Those who have a risk of heart disease, use of pacemaker, epilepsy, transient ischemic attack, stroke or similar nervous disorders and any similar health problems,
* Those with psychiatric, cardiac, pulmonary diseases, pregnant women, those who use drugs that affect the heart rate and blood pressure, those with systemic, neuroplastic, inflammation disorders, those with structural back anomalies, and those who have had lumbar disc herniation complications will not be included in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: During the research process, the participants will divide into 2 groups, then data will collect. Group 1 includes individuals with or without ankle sprain. These are individuals who do not have a history of injury from sprains and are not seeking treatment for similar reasons. Group 2 consisted of participants who have at least one sprained ankle injury/injury at least 2 months ago and who were seeking treatment in the past or on an ongoing basis.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Cumberland Ankle Instabililty Tool (CAIT) | two weeks
  CAIT is a very simple, reliable, and valid measurement tool that is used without comparing with the contralateral ankle, which consists of 9 questions and is scored between 0 and 30, developed by Hiller and her colleagues in 2006 to measure the severity of functional ankle instability. Low scores of the participants indicate poor ankle stability, while high scores indicate good ankle stability .

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Atalay, Md. Phd., Principal Investigator — Department of Sport Medicine, Eskişehir Osmangazi University
Locations (1):
- Eskişehir Technical University, Eskişehir, Tepebaşı, Turkey (Türkiye)

REFERENCES:
- [Derived] Mercanoglu AO, Kacoglu C, Atalay E. Cross-Cultural Adaptation and Cutoff Score Determination of the Turkish Version of the Cumberland Ankle Instability Tool in Recreationally Active Individuals. Orthop J Sports Med. 2025 Aug 19;13(8):23259671251358407. doi: 10.1177/23259671251358407. eCollection 2025 Aug. PMID 40843095